CLINICAL TRIAL: NCT06619483
Title: A Randomized, Single-blind, Placebo-controlled, Single Dose Escalation Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BAY 3018250 in Chinese Healthy Participants
Brief Title: A Study to Learn How Safe BAY3018250 is, How it Moves Into, Through and Out of the Body, and How it Affects the Body in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22491
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Acute Venous and Arterial Thrombotic and Thromboembolic Events; Healthy Volunteers
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAY3018250 Dose 1 (Experimental): Participants will receive BAY3018250 Dose 1.
  Interventions: Drug: BAY3018250 Dose 1
- BAY3018250 Dose 2 (Experimental): Participants will receive BAY3018250 Dose 2.
  Interventions: Drug: BAY3018250 Dose 2
- Placebo (Placebo Comparator): Participants will receive the matching placebo to BAY3018250.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY3018250 Dose 1 — Single dose
  Arms: BAY3018250 Dose 1
Drug: Placebo — Matching placebo to BAY3018250
  Arms: Placebo
Drug: BAY3018250 Dose 2 — Single dose
  Arms: BAY3018250 Dose 2

SUMMARY:
Researchers are looking for a better way to treat people who have acute venous and arterial thrombotic and thromboembolic events.

Acute venous and arterial thrombotic and thromboembolic events refer to blood clots that form and cause blockages in blood vessels that may cause serious complications.

The study treatment BAY3018250 is under development to treat acute venous and arterial thrombotic and thromboembolic events. It works by dissolving blood clots.

In this study, participants will be healthy and will not benefit from BAY3018250. However, the study will provide information about how to test BAY3018250 in future studies of people with acute venous and arterial thrombotic and thromboembolic events.

The results of this study will help in the future development of BAY3018250 as a treatment option for participants with acute venous and arterial thrombotic and thromboembolic events. It will also help in learning more about the drug when given to Chinese participants and helps in involving Chinese sites in clinical trials, to obtain approval for BAY3018250 in China.

The main purpose of this study is to check if BAY3018250 is safe for further testing.

For this, researchers will study the number and severity of medical problems participants have after receiving different amounts of BAY3018250. These medical problems are also known as adverse events. Doctors keep track of all medical problems that happen in studies, even if they do not think they might be related to the study treatment.

In this study, there will be two groups. In each group, participants will be randomly assigned to receive a single dose of either BAY3018250 or placebo as an infusion into a vein, on Day 1. A placebo looks like a study drug but does not have any medicine in it.

In the first group, participants will receive a low dose of BAY3018250. If researchers consider this dose to be safe, the next group will receive a higher dose.

Each participant will be in the study for around 14 weeks, which includes:

a visit to the clinic within 21 days before taking any treatment to confirm if the participant can take part in the study

a hospital stay for around 7 days, during which participants will take their assigned treatment and have blood samples taken to check for drug levels

five follow-ups on Day 10, Day 14, Day 28, Day 42, and Day 75. The last follow-up might be done by phone

During the study, the doctors and their study team will:

collect blood samples from the participants to measure the levels of the study drug given

check participants' health by performing blood and urine tests, measuring the blood pressure, pulse rate and body temperature, and checking heart health using an electrocardiogram (ECG)

ask the participants questions about how they are feeling and what adverse events they are having

As this study is conducted in healthy participants who will not benefit from the treatment, access to the treatment after the study is not planned.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age (both inclusive) at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory test and 12-lead Electrocardiogram (ECG).
* Race: Chinese
* Body mass index (BMI) within the range above or equal to 18.0 to below or equal to 27.9 kg/m*2 at screening.
* Body weight equal or above 55 kg
* Male or postmenopausal or hysterectomized female participants Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent

Exclusion Criteria:

* Increased bleeding risk: known coagulation disorders (e.g., von Willebrand's disease, hemophilia), periodontitis, symptomatic hemorrhoids, acute gastritis, peptic ulcer, or similar diseases with tendency to lead to bleedings, known sensitivity to common causes of bleeding (e.g., nasal, etc.), or history of hemorrhage and gastrointestinal ulceration within 6 months prior to the screening visit.
* Family history of sudden death of unknown reason.
* Family history of hereditary or not explainable bleeding disorders.
* History of thrombosis or family history of hereditary or not explainable diseases with increased risk for thrombosis or thromboembolic events.
* Tendency of easy bruising.
* Use of systemic or topical medicines or substances which oppose the study objectives or which might influence them, e.g. acetylic salicylic acid, heparin, or other Nonsteroidal anti-inflammatory drugs (NSAIDS) or anti-coagulant within 2 weeks or 5 half-lives (whichever is longer) prior to study drug administration or intended during the study.
* Excluded therapies (e.g., physiotherapy, acupuncture, etc.) within 1 week before study intervention administration.
* Platelets out of reference range.
* Activated partial thromboplastin time (aPTT) or prothrombin time (PT) above the upper normal or below 0.5-fold of the lower normal reference range.
* Positive fecal occult blood test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Number of participants who experienced treatment-emergent adverse events (TEAEs) and drug-related TEAEs after administration of BAY3018250 | Administration of study intervention until last follow-up visit (approximately 75 days)

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of BAY3018250 | Pre-dose until Day 42
Area Under the Curve (AUC) of BAY3018250 | Pre-dose until Day 42
  If AUC cannot be determined reliably in all participants, AUC(0-tlast) will be used instead.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou University of TCM, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/22491